CLINICAL TRIAL: NCT00991926
Title: Evaluation of Baseline and Stimulated GH/IGF-1 AXIS in Obese Subjects in Treatment With Orlistat
Brief Title: Growth Factor/Insulin-like Growth Factor (GH/IGF)-1 Axis in Obese Subjects in Treatment With Orlistat
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Annamaria Colao, Dept of Moll Clin Endocrinol Oncol, University Federico II of Naples
Other Study IDs: NeuroendoUnit-12
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Obesity
Keywords: obesity; GH/IGF-1 axis; postprandial NEFA
MeSH Terms: conditions — Obesity | interventions — Orlistat

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- orlistat plus normo-caloric diet: 10 subjects received normo-caloric diet plus + orlistat (Xenical, Roche, UK) at a dose of 120 mg tid. The duration of follow-up was 10 days
  Interventions: Drug: Orlistat; Other: normo-caloric diet
- normo-caloric diet: 10 subjects received normo-caloric diet without the additional treatment. The duration of follow-up was 10 days
  Interventions: Other: normo-caloric diet

INTERVENTIONS:
Drug: Orlistat — orlistat (Xenical, Roche, UK)120 mg tid
  Other Names: gastrointestinal lipase inhibitor
  Groups: orlistat plus normo-caloric diet
Other: normo-caloric diet — Food intake and dietary history were assessed by a skilled dietitian who used a computer-assisted interview (Winfood 1.5, Medimatica srl, Martinsicuro, Italy)

SUMMARY:
The beneficial effects on plasma lipids of Orlistat, a selective gastrointestinal lipase inhibitor, are largely independent of weight loss, and might include differential effects plasma non-esterified fatty acid (NEFA). Apart from their well-known effects on insulin resistance pathogenesis, elevated NEFA levels probably play also the most important role at peripheral levels in the pathogenesis of Growth Hormone (GH) insufficiency in obesity. Aim of this observational, mono-centre, randomized, simple-blind, cross-over study is to verify if the short-term treatment with Orlistat may results in decline in NEFA circulating levels when used in conjunction with low-fat diet and if this effect may restore the endogenous activity of GH/ Insulin-like growth factor (IGF)-1 axis, in the context of GH regulation of lipoprotein metabolism, thus adding a further benefit of Orlistat in obesity cross-linked neuroendocrine and metabolic dearrangement.

DETAILED DESCRIPTION:
Subjects:

Twenty obese postmenopausal women (age: 53.6±6.2; BMI: 34.1±4.0. Subjects were recruited, evaluated, and monitored at the Endocrinology Unit of the Department of Molecular and Clinical Endocrinology and Oncology. Before starting the study, all subjects underwent an initial screening assessment including a medical history, physical examination, laboratory parameters, and body weight.

Treatment protocol:

At study entry plasma samples were obtained for fasting plasma glucose, insulin, lipaemia (total, HDL and LDL cholesterol, tryglycerides), GH, IGF-1, and IGFBP-3. The subjects were randomized in two groups of treatment: 10 subjects received normo-caloric diet plus + orlistat (Xenical, Roche, UK) at a dose of 120 mg tid; 10 subjects received normo-caloric diet without the additional treatment. The duration of follow-up was 10 days for each treatment period, without any wash-out between the two periods. Each patient has been assigned to each group. Dynamic testing performed at the end of each period were the following: glucose, and insulin after an OGTT; GH after GHRH + arginine (GHRH+ARG); post-prandial lipaemia after a standard fat-rich meal. During the study period, the subjects maintained their usual pattern of physical activity. Subjects and investigators remained unaware of laboratory results until the end of the study.

Methods

At baseline and at the end of each period of treatment, the following parameters were also measured:

1. Anthropometric measurements, performed with the subjects wearing only underwear without shoes. Standing height was measured to the nearest cm using a wall-mounted stadiometer. Body weight was determined to the nearest 50 g using a calibrated balance beam scale. Body mass Index (BMI) was calculated as weight (kg) divided by height squared (m2) and used as an index for obesity. Measurements of the waist circumference, a measure of adipose tissue distribution and cardiovascular disease risk were taken at the mid-point between umbilicus and xiphoid.
2. Body composition was determined by conventional Bioelectrical Impedance Analysis (BIA) and by Impedance Vector Analysis (BIVA). Resistance (R) and reactance (Xc) were measured by a single investigator with a single-frequency 50 kHz bioelectrical impedance analyzer (BIA 101 RJL, Akern Bioresearch, Firenze, Italy) according to the standard tetrapolar technique. All evaluations were performed by the same operator blind in respect to subjects treatment.
3. Blood samples were obtained between 08:00 h and 09:00 h from antecubital vein after an overnight fast, with the patient in the resting position. Blood samples for hormonal determination were promptly centrifuged, and serum separated and stored at -20 C until assay. Blood glucose levels were determined by the glucose oxidase method immediately after the OGTT. The OGTT was performed using 75 g dextrose. Blood samples were obtained at 0, 30, 60, 90, 20, 150, and 180 minutes for plasma glucose and insulin measurements. The normal glycemic response to the OGTT was defined according to the criteria of the Expert Committee on the Diagnosis and Classification of Diabetes Mellitus . Total and HDL-cholesterol, and triglyceride concentrations were assayed in plasma by enzymatic colorimetric methods (Roche Molecular Biochemicals) on an autoanalyzer Cobas Mira (ABX Diagnostics). LDL-cholesterol was calculated using Friedewald formula. Changes in lipid profile was also analyzed by calculating the total/HDL cholesterol ratio. Plasma NEFA concentrations were analyzed by the enzymatic colorimetric method (Wako Chemicals). Serum insulin and c-peptide were measured by a solid-phase chemiluminescent enzyme immunoassay using commercially available kits (Immunolite Diagnostic Products Co, Los Angeles, CA, USA). The sensitivity of the assay were 0.1 and 0.3 ng/mL. The intra- and interassay coefficients of variations (CVs.) were 2.2 and 5.8%, respectively for insulin and 6.3 and 8.8%, respectively for c-peptide.

The GHRH (1-29, Geref, Serono, Rome, Italy)+ ARG (arginine hydrochloride, Salf, Bergamo, Italy) was performed. The GH response after ARG+GHRH was classified as deficient (GHD) when the GH peak was <4.2 µg/L and sufficient (GHS) when the GH peak was >4.2 µg/L. Serum GH levels were measured by immunoradiometric assay (IRMA) using commercially available kits (HGH-CTK-IRMA, Sorin, Saluggia, Italy). The sensitivity of the assay was 0.02 µg/L. The intra- and interassay coefficients of variations (CVs.) were 4.5 and 7.9%, respectively. Circulating IGF-I levels measured by IRMA after ethanol extraction using Diagnostic System Laboratories Inc. (Webster, Texas, USA). The normal ranges in 31-40, 41-50 and 51-60 yr old women were 100-390, 96-288, 90-250 µg/l, respectively. The sensitivity of the assay was 0.8 µg/l. The intra-assay CVs were 3.4, 3.0 and 1.5% for low, medium and high points of the standard curve, respectively. The inter-assay CVs were 8.2, 1.5 and 3.7% for low, medium and high points of the standard curve. For the purpose of this study, IGF-I levels were classified as normal when higher than -2 SD and deficient when it was lower than -2 SD. The IGFBP-3 assay had a sensitivity of 0•04 ng/l; the normal range for an adult female population of the same age range of our study population was 2.7-5.6 mg/L. The values for the molecular mass of IGF-I and IGFBP-3 used for the calculation were 7.649 kDa and 28.5 kDa, respectively.25 Post-prandial lipaemia was evaluated in the morning, after ≥ 12 h fasting, and over the 8 h following the standard meal (at 2, 4, 6 and 8) h. The standard meal consisted of a potato gateau (a pie made of mashed potato, whole milk, egg, cheese, ham and butter) which was consumed in 15-20 min. The meal, which provided 4090 kJ, was composed of 34% carbohydrates, 51% fat (34% saturated fat) and 15% protein.

ELIGIBILITY:
Inclusion Criteria:

* women
* post-menopausal age
* class I-II obesity
* normal thyroid, liver, and kidney function

Exclusion Criteria:

* type 2 diabetes mellitus
* use of hypolipaemic agents

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: nondiabetic obese post-menopausal women
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2006-12; Primary Completion 2006-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
GH/IGF-1 axis (GH at baseline and after GHRH+Arg; IGF-1, IGFBP3, IGF-1/IGFBP3 ratio) | 20 days

SECONDARY OUTCOMES:
fasting lipaemia (total, HDL and LDL cholesterol, tryglycerides, NEFA, total/HDL cholesterol ratio | 20 days
post-prandial lipaemia (total, HDL and LDL cholesterol, tryglycerides, NEFA) | 20 days
Antropometric indexes: Body mass index (BMI), waist circumference | 20 days
glucose metabolism: OGTT, Insulin resistance (HOMA-R - homeostasis model assessment of insulin resistance) index, Insulin Sensitivity Index (ISI) | 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Colao, MD, PhD, Principal Investigator — Department of Molecular and Clinical Endocrinology and Oncology Federico II University of Naples

REFERENCES:
- [Derived] Di Somma C, Rivellese A, Pizza G, Patti L, De Rosa A, Cipriano P, Nedi V, Rossi A, Lombardi G, Colao A, Savastano S. Effects of short-term treatment with orlistat on growth hormone/insulin-like growth factor-I axis in obese post-menopausal women. J Endocrinol Invest. 2011 Feb;34(2):90-6. doi: 10.1007/BF03347036. PMID 21502796